CLINICAL TRIAL: NCT04663243
Title: Effectiveness of Thinking Healthy Program for Prevention of Antenatal Depression to Improve Maternal Health, Pakistan
Brief Title: Effectiveness of Thinking Healthy Program for Prevention of Antenatal Depression
Acronym: PAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Punjab (Other)
Responsible Party: Principal Investigator, Quratulain Ahsan, Principal Investigator, University of the Punjab
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: THP in clinical settings
Record Dates: First submitted 2020-10-30; First posted 2020-12-10 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2021-09

CONDITIONS: Post Partum Depression
Keywords: Antenatal depression; psychosocial factors; Thinking Healthy Program
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: Quasi experimental study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Quasi experimental study (Experimental): Before intervention and after intervention comparison
  Interventions: Behavioral: Thinking healthy Program sessions designed for antenatal period

INTERVENTIONS:
Behavioral: Thinking healthy Program sessions designed for antenatal period — Low line psychosocial intervention based on the principles of Cognitive Behavior Therapy (CBT), designed for non-specialist will be applied for expectant women experiencing depression during mid to late-pregnancy. It uses the core principles and strategies of the Thinking Healthy Program (THP). Four core sessions and two booster sessions will be applied, designed for antenatal period to prevent antenatal and post partum depression.
  Other Names: Psychoeducation

SUMMARY:
The trial is to evaluate the effect of an evidence-informed, depression focused early prenatal prevention intervention at six weeks' postpartum. Secondary objective is to explore demographical and psychosocial factors responsible for development of prenatal and postpartum depression. Investigator will also examine the potential mediators of depression and the effect of intervention on depression and its related factors i.e. marital relationship, social support, empowerment and history of intimate partner violence. Pregnant women coming for their antenatal visits to the Sheikh Zayed Hospital (SZH), a public facility in Lahore, Pakistan, will be screened for eligibility. Eligible women will be 24-26 weeks pregnancy who will be assessed as having mild to moderate levels of depression [i.e., score ≥10 on Personal Health Care Questionnaire (PHQ-9)] validated in Pakistan for the use of non-specialist.

DETAILED DESCRIPTION:
The present study aims to evaluate the effectiveness of evidence informed, depression focused early prenatal prevention intervention in pregnant women at six weeks' postpartum. Investigator hypothesize that women with subclinical to clinical levels of prenatal depression to the intervention will result in fewer cases of depression (mild to moderate) at six weeks' postpartum. The primary objective of the trial is to evaluate the effect of an evidence-informed, depression focused early prenatal prevention intervention at six weeks' postpartum. Secondary objective is to explore demographical and psychosocial factors responsible for development of prenatal and postpartum depression. We will also examine the potential mediators of depression and the effect of intervention on depression and its related factors i.e. marital relationship, social support, empowerment and history of intimate partner violence. Pregnant women coming for their antenatal visits to the Sheikh Zayed Hospital (SZH), a public facility in Lahore, Pakistan, will be screened for eligibility. Eligible women will be 24-26 weeks pregnancy who will be assessed as having mild to moderate levels of depression [i.e., score ≥10 on Personal Health Care Questionnaire (PHQ-9)] validated in Pakistan for the use of non-specialist.

An intervention thinking Healthy Program (THP) will be done in which Investigator will enroll up to twenty (20) pregnant women. Low line psychosocial intervention based on the principles of Cognitive Behavior Therapy (CBT), designed for non-specialist will be applied for expectant women experiencing depression during mid to late-pregnancy. It uses the core principles and strategies of the Thinking Healthy Program (THP), an evidence-based psychosocial intervention for mothers experiencing perinatal depression, including empathetic listening, thought challenging, behavior activation, family involvement, and problem management. Additionally, stress management skills such as breathing exercises are incorporated. Culturally relevant customized illustrations are used for guided discovery, behavior activation, stress management, and to convey key health messages. The intervention is a series of one-on-one sessions, complemented by take home exercises. Before and after intervention comparison will be made to find out the efficacy of intervention. The data will be collected at one site: Sheikh Zayed Hospital, a public tertiary care facility in Lahore, Pakistan. It will take six months for data collection.

ELIGIBILITY:
Inclusion Criteria:

* Women with 24-26 weeks pregnancy.
* Women assessed as having mild to moderate levels of depression [i.e., score ≥10 on Personal Health Care Questionnaire (PHQ-9)] tool validated in Pakistan for the use of non-specialist.

Exclusion Criteria:

* Women having depression severe depression [i.e., score ≥20 on Personal Health Care Questionnaire (PHQ-9)]
* Women will be diagnosed serious medical condition requiring inpatient or outpatient treatment,
* Pregnancy-related illness (except for common conditions, such as anaemia)
* Any physical or learning disability or other form of psychosis
* Women younger than 18 and greater than 45 years will also be excluded.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Women with 24-26 weeks pregnancy who will be assessed as having mild to moderate levels of depression [i.e., score ≥10 on Personal Health Care Questionnaire (PHQ-9)] tool validated in Pakistan for the use of non-specialist.
Enrollment: 22 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2021-01-29 (Actual); Study Completion 2021-04-29 (Actual)

PRIMARY OUTCOMES:
Assessment of antenatal depression | Five months
  Screening of patients with antenatal depression using PHQ-9 tool for calculation of percentage(%) of depressive women in pregnancy before 6 sessions of Thinking Healthy Program
Assessment of postpartum depression after 6 sessions of Thinking Healthy Program | After delivery to 6 weeks (puerperium period)
  Screening of patients with post depression using PHQ-9 tool for calculation of percentage(%) of depressive women in postpartum period

CONTACTS AND LOCATIONS:
Overall Officials: Abid Malik, PhD, Study Chair — Human Development Research Foundation, Pakistan
Locations (1):
- Sheikh Zayed Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
The primary objective of the trial is to evaluate the effect of an evidence-informed, depression focused early prenatal prevention intervention at six weeks' postpartum. Secondary objective is to explore demographical and psychosocial factors responsible for development of prenatal and postpartum depression. Pregnant women coming for their antenatal visits to the Sheikh Zayed Hospital (SZH), a public facility in Lahore, Pakistan, will be screened for eligibility. Eligible women will be 24-26 weeks pregnancy who will be assessed as having mild to moderate levels of depression [i.e., score ≥10 on Personal Health Care Questionnaire (PHQ-9)].
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 30-3-2021
Access Criteria: Data will be available in the form of publication, after the acceptance of paper.

REFERENCES:
- [Derived] Ahsan Q, Saleem J, Ishaq M, Zakar R, Abbas S, Shahzad R, Khan SM, Fischer F. Determinant factors and coping strategies for depression among pregnant women: an intervention-based qualitative study in Lahore, Pakistan. BMC Psychiatry. 2024 Nov 19;24(1):829. doi: 10.1186/s12888-024-06280-3. PMID 39563299

DOCUMENTS (2):
  • Study Protocol (2020-06-23): https://cdn.clinicaltrials.gov/large-docs/43/NCT04663243/Prot_000.pdf
  • Informed Consent Form (2020-03-13): https://cdn.clinicaltrials.gov/large-docs/43/NCT04663243/ICF_001.pdf